CLINICAL TRIAL: NCT06404671
Title: Timing of Surgery After Neoadjuvant Chemotherapy for Advanced Ovarian Cancer: A Randomized Clinical Trial for Early Versus Delayed Interval Cytoreductive Surgery
Brief Title: Timing of Surgery After Neoadjuvant Chemotherapy for Advanced Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGOU 1
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Epithelial Cancer
Keywords: high grade serous; advanced primary ovarian cancer; interval cytoreduction
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed interval cytoreduction surgery (DICS) (Experimental): delayed interval cytoreduction surgery after six courses of intravenous carboplatin and paclitaxel every 3 weeks
  Interventions: Procedure: Delayed interval cytoreductive surgery (DICS)
- Early interval cytoreduction surgery (EICS) (Active Comparator): Early interval cytoreduction surgery after three courses of intravenous carboplatin and paclitaxel every 3 weeks
  Interventions: Procedure: Early interval cytoreductive surgery (EICS)

INTERVENTIONS:
Procedure: Delayed interval cytoreductive surgery (DICS) — patients will receive six courses of intravenous carboplatin and paclitaxel every 3 weeks, followed by delayed interval cytoreductive surgery (DICS) within 6 weeks of the last cycle of chemotherapy. After DICS, patients will be assessed for the need or not for further adjuvant chemotherapy.
  chemotherapy regimen:
  * Paclitaxel at 175 mg/m² + carboplatin area under the curve (AUC) 5-6 every 3 weeks.
  * Paclitaxel at 60 mg/m² (days 1, 8, and 15), and carboplatin AUC 2 (days 1, 8, and 15) every 3 weeks.
  * Paclitaxel at dense dose 80 mg/m² (days 1, 8, and 15) and carboplatin AUC 5-6 (day 1) every 3 weeks.
  Arms: delayed interval cytoreduction surgery (DICS)
Procedure: Early interval cytoreductive surgery (EICS) — patients will receive three courses of intravenous carboplatin and paclitaxel every 3 weeks, followed by early interval cytoreductive surgery (EICS) within 6 weeks of the last cycle of chemotherapy. After EICS, patients will receive adjuvant three courses of intravenous carboplatin and paclitaxel every 3 weeks, then will be assessed for the need or not for further adjuvant chemotherapy.
  chemotherapy regimen:
  * Paclitaxel at 175 mg/m² + carboplatin area under the curve (AUC) 5-6 every 3 weeks.
  * Paclitaxel at 60 mg/m² (days 1, 8, and 15), and carboplatin AUC 2 (days 1, 8, and 15) every 3 weeks.
  * Paclitaxel at dense dose 80 mg/m² (days 1, 8, and 15) and carboplatin AUC 5-6 (day 1) every 3 weeks.
  Arms: Early interval cytoreduction surgery (EICS)

SUMMARY:
Ovarian cancer is among the top five primary causes of cancer-related mortality in women. Most ovarian malignant tumours originate from epithelial cells The majority of patients typically have advanced-stage tumours at diagnosis. When complete surgery with no macroscopic visible disease is not feasible due to both the spread of the disease and the patient's general condition, neoadjuvant chemotherapy (NACT) of 3 cycles followed by interval cytoreductive surgery (ICS) or final cytoreductive surgery (FCS) after 6 cycles of NACT followed or not by adjuvant chemotherapy can be offered, with similar overall survival. In our centre, due to logistics, disease, or patient factors, many patients may receive more than 3 cycles of NACT before ICS. Therefore, this randomized controlled trial aims to evaluate the survival benefit of different timings of ICS after 3 or 6 cycles of NACT in patients not eligible for upfront cytoreductive surgery (UCS).

ELIGIBILITY:
Inclusion Criteria:

1. Female Patients aged 18 to 75 years.
2. International Federation of Gynecology and Obstetrics (FIGO) stage IIIB-IV unsuitable for UCS.
3. Histologically confirmed high-grade serous (HGS) ovarian, fallopian tube, or primary peritoneal carcinoma.
4. ECOG performance status: 0 or 1.
5. Resectable disease by laparoscopic assessment after 3 cycles of NACT.
6. Adequate haematology, bone marrow, respiratory, hepatic, cardiac and renal functions.
7. Estimated life expectancy of > 3 months according to Age-adjusted Charlston Co-morbidity Index (ACCI), included patients should have a low or intermediate comorbidity score; ACCI 0-3.

Exclusion Criteria:

1. Metastatic ovarian carcinoma.
2. Patients with primary ovarian carcinoma other than high-grade serous (low-grade serous, endometrioid, mucinous, clear cell, and non-epithelial ovarian carcinoma).
3. Presence of pregnancy or breast-feeding.
4. History of other invasive malignancies in the previous 5 years.
5. History of a recent < 6 month cerebrovascular accident.
6. Uncontrolled systemic disease or contraindication to chemotherapy.
7. Progressive disease on NACT.
8. Worsening Eastern Cooperative Oncology Group (ECOG) Performance Status (ECOG 2-4).
9. Severe comorbidities (ACCI >= 4)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 5years
  PFS will be defined as the time to recurrence/progression, or the date of death. Disease recurrence/ progression is defined as an increase in cancer antigen 125 (CA 125) levels or evidence of recurrence by imaging and/or histology.
Overall survival (OS) | up to 5 years
  OS will be defined as the time until the patient's death from any cause. The time to event occurrence will be calculated from the time of randomization until the event of interest.

SECONDARY OUTCOMES:
Operative peritoneal cancer index (PCI) assessment | 3-6 months
  pre- and post-operative PCI
Complete resection rate | 3-6 months
  proportion of patients without macroscopically visible disease according to residual (R), patients will have R0 if no macroscopic residual, R1 if the residual is ≤10 mm, and R2 if the residual is > 10 mm.
Surgical complexity scoring (low, intermediate, or high) | 3-6 months
  assessment of complexity score of during surgery
Post-operative morbidity | within 30 days of surgery
  Post-operative morbidity according to the Clavien-Dindo classification (CDC), i.e., proportion of severe complications (CDC grade 3-5) within 30 days of surgery.
Pathological complete chemotherapy response score (CRS 3) | 3-6 months
  Pathological complete chemotherapy response score (CRS 3) in the pathology specimen
The total number of chemotherapy cycles administered | 8 months
  The total number of chemotherapy cycles administered (NACT + adjuvant cycles).
Tumour recurrence and death | Up to 5 years
  Proportion of patients who had recurrence or died in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Elshatby Maternity University Hospital, Alexandria, Egypt